CLINICAL TRIAL: NCT04241913
Title: A Randomized Controlled Trial to Improve Biobehavioral Regulation Among High-Adversity Mothers and Young Children
Brief Title: Mom Power With High-Adversity Mothers and Children
Acronym: MPHAMC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and pandemic-related mitigation strategies, we were forced to alter procedures prior to the enrolling of participants into this trial. We will submit a new protocol for our adapted trial, launching at a later date.
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Gray, Assistant Professor of Psychology, Clinical Professor of Psychiatry & Behavioral Sciences, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-2012; 1K23MH119047-01 (NIH)
Record Dates: First submitted 2020-01-10; First posted 2020-01-27 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Self-regulation; Respiratory Sinus Arrhythmia
Keywords: biobehavioral self-regulation; psychopathology; parenting behavior
MeSH Terms: conditions — Self-Control; Arrhythmia, Sinus

STUDY DESIGN:
Intervention Model Description: There are two arms: an experimental group receiving the Mom Power group intervention over 10 weeks, and a wait list control group. Treatment delivery will be consistent with the Mom Power manual. The waitlist control group will be offered to participate in the intervention following the trial period.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment group receives the 10-week, group-based Mom Power intervention; intervention is provided to both mothers and children by trained providers. Treatment delivery will be consistent with the Mom Power manual.
  Interventions: Behavioral: Mom Power Intervention
- Waitlist control (No Intervention): Participants randomized to waitlist control will not receive treatment during the experimental period; they will be offered treatment following completion of post- assessments.

INTERVENTIONS:
Behavioral: Mom Power Intervention — Mom Power is a 10-week therapeutic intervention for at-risk families that incorporates elements of several evidence based practices. It combines didactic material with mindbody self-care skills and in vivo practice to improve the quality of attachment between parent and child, and to reduce the psychopathology of at-risk parents. The child team component provides each child with one-on-one care focusing on meeting the child's social-emotional needs and providing attachment-related experiences within a developmental framework.
  Arms: Treatment

SUMMARY:
This study will evaluate whether the intervention, Mom Power, improves the self-regulation of mothers with a history of trauma and their children. The central hypothesis is that the intervention will shift behavioral and physiological self-regulation in mothers, children, and dyads to mitigate psychopathology risk.

DETAILED DESCRIPTION:
Adverse childhood experiences (ACEs) are significant risk factors for psychopathology across the lifespan - risks that extend to the next generation, likely transmitted through both biological and behavioral pathways. Biobehavioral self-regulation and parenting are key candidates for transmission and potential points of intervention. However, nearly all intervention research takes a one-generation approach, measuring outcomes in the individual adult or child in treatment. Additionally, very little research has examined biomarkers of self-regulation in parents or children following treatment, and no known research has examined these processes in parents and young children simultaneously across treatment to explore bidirectional effects. There is a critical need to specify targets of two-generation interventions among high-adversity families to decrease intergenerational transmission of mental illness. The objective of this RCT is to determine whether Mom Power, an evidence-based two generation intervention for mothers with histories of trauma, enhances physiological and behavioral self-regulation in mothers and young children, testing mechanisms and examining bidirectional effects. The central hypothesis is that the intervention will shift behavioral and physiological (Respiratory Sinus Arrhythmia) self-regulation in mothers, children, and dyads to mitigate psychopathology risk. Three specific aims are proposed: 1) Examine intervention effects on children's biobehavioral self-regulation and psychopathology; 2) Examine intervention effects on mothers' biobehavioral self-regulation, psychopathology, and parenting behavior; and 3) Examine intergenerational change processes, including shifts in dyadic physiological and behavioral synchrony as well as bidirectional influences between mother and child self-regulation.

ELIGIBILITY:
Participants in this study must include a mother-child dyad. There is inclusion and exclusion criteria for both mother and child.

Inclusion Criteria:

* For moms: Mothers must be female, the biological mother, have an ACE score of 3 or more, speak English, and be 18 years or older.
* For children: Children must be between the ages of 2 and 5.

Exclusion Criteria:

* For mothers: No pacemaker or self-reported heart condition; no active maternal substance abuse or psychosis on screeners (Brown & Rounds, 1995; Degenhardt, Hall, Korten, & Jablensky, 2005).
* For children: No parent report of diagnosis of autism or global development delay, no parent report of pacemaker or heart condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Child participants can be male or female. Recruited parent must be biological mother due to interest in intergenerational patterns and concerns about heritability of the primary outcome.
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Child RSA | Within 6 weeks of treatment group completion; approximately 4 months
  Child self-regulation will be assessed physiologically with RSA baseline and RSA change during a parent-child dyadic task (Skowron et al., 2013); derived from electrocardiogram (ECG) collected using Mindware Technologies ambulatory mobile recorders during 1) 2-minute resting baseline; 2) a dyadic interaction task. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify RSA within frequency bandwidths associated with respiration (.15-.40 for mothers; .24-1.04 for children), processed in 1-minute epochs averaged across tasks, and log-transformed.
Parent RSA | Within 6 weeks of treatment group completion; approximately 4 months
  Parent self-regulation will be assessed physiologically with RSA baseline and RSA change during a parent-child dyadic task (Skowron et al., 2013); derived from electrocardiogram (ECG) collected using Mindware Technologies ambulatory mobile recorders during 1) 2-minute resting baseline; 2) a dyadic interaction task. ECG signals will be synchronized at acquisition with video and processed offline using Mindware software; research assistants will visually inspect for missing or erroneously identified R-peaks. Using spectral analysis of interbeat intervals, high-frequency heart rate variability will be extracted to quantify RSA within frequency bandwidths associated with respiration (.15-.40 for mothers; .24-1.04 for children), processed in 1-minute epochs averaged across tasks, and log-transformed.

SECONDARY OUTCOMES:
Child Behavior - parent report | Within 6 weeks of treatment group completion; approximately 4 months
  Child Behavior problems will be assessed via Total Score on parent report with the Child Behavior Checklist; higher scores indicate higher behavior problems (T score is a standardized score with a mean of 50).
Child Behavior - teacher report | Within 6 weeks of treatment group completion; approximately 4 months
  Child Behavior problems will be assessed via teacher report with the Teacher Report Form; Achenbach & Rescorla, 2000. Higher scores indicate higher behavior problems (T score is a standardized score with a mean of 50).
Dyadic synchrony - physiological | Within 6 weeks of treatment group completion; approximately 4 months
  Dyadic synchrony will be assessed using EKG (derived from maternal and child RSA, as described above)
Dyadic synchrony - observational | Within 6 weeks of treatment group completion; approximately 4 months
  Dyadic synchrony will be assessed observationally with the Coding Interactive Behavior (CIB) measure.
Parent psychopathology | Within 6 weeks of treatment group completion; approximately 4 months
  Parents will report on their own depression symptoms (Patient Health Questionnaire-9 and Posttraumatic Checklist - 5); individual scales will be z-scored and summed, with higher values reflecting higher levels of psychopathology
Parent emotion regulation | Within 6 weeks of treatment group completion; approximately 4 months
  Parents will report on their own emotion regulation using the difficulties in emotion regulation (DERS; range: 36-180); higher scores reflect more difficulties with emotion regulation.
Sensitive parenting behavior | Within 6 weeks of treatment group completion; approximately 4 months
  Observational data derived from parent-child interactions will be examined, coding using the Coding Interactive Behavior measure (CIB). Higher scores reflect more sensitivity.
Parent self-efficacy | Within 6 weeks of treatment group completion; approximately 4 months
  Parents will report on their own parenting efficacy using the Parent Sense of Competence scale; range: 17-102, higher scores reflect more self-efficacy
Parenting behavior | Within 6 weeks of treatment group completion; approximately 4 months
  Parents will report on their own parenting behavior using the Conflict Tactic Scales - Parent Child (CTS-PC); range: 0-240, higher values reflect harsher parenting
Parent mental representation | Within 6 weeks of treatment group completion; approximately 4 months
  Parents will complete an abbreviated version of the Working Model of the Child Interview; interviews will be coded into 3 categories, and it is hypothesized that proportion of "balanced" representations will be higher post-treatment.
Child Behavioral Self-Regulation, observational | Within 6 weeks of treatment group completion; approximately 4 months
  Child self-regulation will be assessed behaviorally using observation (Preschool Self-Regulation Assessment); children's behavior will be observed during 6 tasks, and codes z-scored and summed; higher scores reflect higher effortful control/executive function
Child Behavioral Self-Regulation, parent report | Within 6 weeks of treatment group completion; approximately 4 months
  Child self-regulation will also be assessed by parent-report (Social Competence Scale - Emotion Regulation); range: 0-48; higher scores reflect higher self-regulation

OTHER OUTCOMES:
Maternal social support | Within 6 weeks of treatment group completion; approximately 4 months
  Mothers will report on social support (Multidimensional Scale of Perceived Social Support); range: 12-84; higher scores reflect higher perceived support.
Perceived stress | Within 6 weeks of treatment group completion; approximately 4 months
  Mothers will report on perceived stress (Perceived Stress Scale-4); range: 0-16; higher scores reflect higher stress

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Gray, PhD, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - Educare New Orleans, New Orleans, Louisiana
  - Kingsley House Early Head Start Preschool, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenblum KL, Muzik M, Morelen DM, Alfafara EA, Miller NM, Waddell RM, Schuster MM, Ribaudo J. A community-based randomized controlled trial of Mom Power parenting intervention for mothers with interpersonal trauma histories and their young children. Arch Womens Ment Health. 2017 Oct;20(5):673-686. doi: 10.1007/s00737-017-0734-9. Epub 2017 Jun 25. PMID 28647759
- See also: Bibliography of Sarah Gray, PhD — https://www.ncbi.nlm.nih.gov/sites/myncbi/sarah.gray.2/bibliography/49443145/public/?sort=date&direction=as